CLINICAL TRIAL: NCT03980795
Title: Resistance and Cardiovascular Exercise for Peritoneal Dialysis Patients: a Randomized Pilot Study for a Parallel Randomized Controlled Trial
Brief Title: Exercise in Peritoneal Dialysis Patients (PDEX)
Acronym: PDEX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Satellite Healthcare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SH107
Record Dates: First submitted 2019-05-29; First posted 2019-06-10 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: Peritoneal Dialysis; Kidney Failure, Chronic
Keywords: exercise; physical function; patient reported outcomes
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded Statistical Analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention (I) group received monthly exercise physiologist consultations, exercise prescription (resistance and aerobic exercise program using exercise bands) and weekly phone calls over 12 weeks.
  Interventions: Other: Exercise Program
- Control (No Intervention): Usual care

INTERVENTIONS:
Other: Exercise Program — Participants met with an exercise physiologist at their monthly center appointment over a 3-month period (4 meetings). The consultations took place either together or separate from or with the dietitian's consultation (depending on appointment logistics). In addition the Exercise Physiologists telephone called each intervention participant on a weekly basis.
  Arms: Intervention

SUMMARY:
Patients with end-stage kidney disease (ESKD) receiving peritoneal dialysis (PD) are physically inactive, resulting in poor physical function and reduced quality of life. The aim of this pilot trial was to test the study feasibility of a combined resistance and cardiovascular exercise program (recruitment and retention rates) and report adherence and adverse events. The intervention (I) group received monthly exercise physiologist consultations, exercise prescription (resistance and aerobic exercise program using exercise bands) and weekly phone calls over 12 weeks. Control (C) group received normal care. Feasibility outcomes were exercise adherence rates and adverse events. Secondary measures included physical function measures and patient-reported outcome measures (PROMs)

DETAILED DESCRIPTION:
Patients with end-stage kidney disease (ESKD) receiving peritoneal dialysis (PD) are physically inactive, resulting in poor physical function and reduced quality of life. Combined resistance and cardiovascular exercise programs have been shown to be successful in hemodialysis patients but studies are limited in PD patients. The primary objectives of this pilot trial was to test the study feasibility of a combined resistance and cardiovascular exercise program (recruitment and retention rates) and report adherence and adverse events. Secondary objectives were to calculate the sample size for detecting differences in the 30 second sit to stand test (STS30) and measure the effect on physical function and patient reported outcome measures (PROMs).

Methods: The 3-month parallel two-arm pilot trial took place in California, USA. All participants were peritoneal dialysis patients in a single center who met inclusion criteria were invited into a randomized controlled trial. Recruitment was through face to face invitation following eligibility requirements. The intervention (I) group received monthly exercise physiologist consultations, exercise prescription (resistance and aerobic exercise program using exercise bands) and weekly phone calls over 12 weeks. Control (C) group received normal care. Feasibility outcomes were exercise adherence rates and adverse events. Secondary physical function measures were change in I compared to the C group in STS30, pinch strength test (PST) and the 8 foot timed up and go test (8TUG). PROMs were measured using the London Evaluation of Illness (LEVIL) instrument. Data collection was not blinded but statistical analysis was blinded.

ELIGIBILITY:
Inclusion Criteria:

* end-stage kidney disease
* receiving peritoneal dialysis for greater than 6 weeks
* approved by the center Medical Director

Exclusion Criteria:

* unable to understand English
* previous major amputations
* unable to ambulate independently
* known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of Study - number of patients safely completing the study | 1 month
  The number of patients safely completing the study relative to the sampling frame
Adherence to exercise - total number of self-reported exercise sessions attempted divided by the total number of exercise sessions prescribed | 3 months
  the total number of self-reported exercise sessions attempted divided by the total number of exercise sessions prescribed

SECONDARY OUTCOMES:
30 second sit to stand test | 3 months
  Requires a participant to stand from a chair as many times as possible in 30 seconds
Pinch Strength Test | 3 months
  consists of three pinch tests: the tip pinch, lateral pinch and palmar pinch. All were performed following the American Society of Hand Therapists' recommendations
Timed Up and Go | 3 months
  the time in seconds it takes an adult to rise from sitting in a standard chair, walk 8 feet, turn, walk back to the chair and sit down using regular footwear

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Schiller, MD, Principal Investigator — Satellite Healthcare
Locations (1):
- Satellite Wellbound Sacramento, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
All feasibility data will be published
Supporting Information: CSR
Time Frame: De-identified data will be available. Results will disseminated through peer reviewed publication.

REFERENCES:
- [Derived] Bennett PN, Hussein WF, Matthews K, West M, Smith E, Reiterman M, Alagadan G, Shragge B, Patel J, Schiller BM. An Exercise Program for Peritoneal Dialysis Patients in the United States: A Feasibility Study. Kidney Med. 2020 Mar 17;2(3):267-275. doi: 10.1016/j.xkme.2020.01.005. eCollection 2020 May-Jun. PMID 32734246